CLINICAL TRIAL: NCT02865486
Title: The Effect of Biopolymer Based Lipid Emulsions on GI Function, GI Peptide Response and Satiation in Healthy Volunteers; a Randomized, Double Blind, Unbalanced Three-way Crossover Study
Brief Title: Digestion of Biopolymer Based Lipid Emulsions
Acronym: BioLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BASEC 2015-00032
Record Dates: First submitted 2016-04-14; First posted 2016-08-12 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Gastric emptying; MRI; lipid emulsions; breath test; GI peptide hormones
MeSH Terms: interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lipid emulsion: visit 2 (Experimental): One of four randomly assigned lipid emulsions
  Interventions: Dietary Supplement: Lipid emulsion
- Lipid emulsion: visit 3 (Experimental): One of four randomly assigned lipid emulsions
  Interventions: Dietary Supplement: Lipid emulsion
- Lipid emulsion: visit 4 (Experimental): One of four randomly assigned lipid emulsions
  Interventions: Dietary Supplement: Lipid emulsion

INTERVENTIONS:
Dietary Supplement: Lipid emulsion — 1 of 4 isovolumetric (200 ml) and isocaloric (380 kcal) lipid emulsions with different acid and shear stability will be ingested on visit 2.
  Arms: Lipid emulsion: visit 2
Dietary Supplement: Lipid emulsion — 1 of 4 isovolumetric (200 ml) and isocaloric (380 kcal) lipid emulsions with different acid and shear stability will be ingested on visit 3.
  Arms: Lipid emulsion: visit 3
Dietary Supplement: Lipid emulsion — 1 of 4 isovolumetric (200 ml) and isocaloric (380 kcal) lipid emulsions with different acid and shear stability will be ingested on visit 4.
  Arms: Lipid emulsion: visit 4

SUMMARY:
In this randomized, double blind, unbalanced three way crossover trial, four lipid emulsions will be assessed on three study days. The lipid emulsions (LEs) have been engineered so that they differ in terms of acid stability, lipid droplet size and fat redispersibility. The investigators hypothesize that the gastric emptying of fat will differ between the lipid emulsions.

An optional study day (visit 5) will be used to assess the degree of lipolysis in Lipid emulsion 5 (LE5) and Lipid emulsion 6 (LE6). This study day is a randomized, single blinded study.

DETAILED DESCRIPTION:
The physical state of fat has been demonstrated to affect the rate of fat digestion. By engineering the physical properties of lipid emulsions the investigators are able to alter characteristics such as acid stability, lipid droplet size and fat redispersibility. These factors have been shown to modulate the physical state of fat in the stomach, the subsequent fat gastric emptying and digestion as well as satiation in healthy subjects. The investigators have recently developed a new series of lipid emulsions based on biopolymers. Preliminary animal studies have shown that these emulsions are able to effect GI physiology including GI peptide hormones and eating behavior. The primary aim of this work is to apply these biopolymer based lipid emulsions in healthy subjects and investigate their impact on fat digestion and satiation. A secondary aim is to develop an image analysis method that can quantify the heterogeneity of fat distribution within gastric content from the MRI data.

The participants (n=17) will be randomized at screening to receive 3 of the 4 lipid emulsions (LE).

On each of the three study days subjects will receive 200 mL of a lipid emulsion. MRI scans will be performed at regular intervals over a period of 3.5 h. Blood samples (for GI peptide hormone analysis) will also be taken at regular intervals until 5 h post LE ingestion. Further, 13C breath test samples will be obtained from participants every 10 min until 5 h post ingestion of LE. Throughout the entire 5 h study period participants will be asked to score their visceral sensation in relation to satiation. Once the technical section of the study is complete the participant will be provided with an ad libitum buffet from which they can consume as much or a little of the food options provided in the buffet.

Optional study day: After the main study is complete and the MRI data has been analyzed the study will be unblinded. This will enable the investigators to optimize an MR imaging and gastric content sampling schedule for LE5 and LE6. The participants (n=17) will be randomized and 10 subjects will then be given the opportunity to participate in the optional study day. The optional study day is single blinded and consists of 1 extra visit and is of a maximum 3 h duration. No bloods, breath test samples or visceral sensation scores will be taken. Subjects will arrive fasted and a nasogastric tube will be positioned. 200 mL of either LE5 or LE6 containing the 13C breath test marker will then be infused. MR imaging will continue at defined intervals until maximum of 3 h. In total five gastric content samples of 5 mL will be taken with the nasogastric tube.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 kg/m²
* Written informed consent

Exclusion Criteria:

* Donated blood within the last 3 months
* History of GI, cardiorespiratory (including arterial
* hypertension), hematologic, renal, atopic, alimentary or psychiatric disorder, panic attacks, diabetes
* Prior abdominal surgery other than uncomplicated appendectomy or hernia repair
* Requiring medication that might alter gut function, including calcium channel blockers, prokinetics, macrolide antibiotics
* Presence of metallic implants, devices or metallic foreign bodies
* Pregnancy and lactation (female participants of child bearing age will receive a pregnancy test prior to study)
* Claustrophobia
* Regular smoking
* A history of drug or alcohol abuse
* A history of food allergies or intolerances
* Uncertainty about the willingness or ability of the participant to comply with the protocol requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The rate of gastric fat volume emptying [ml/h] | up to 210 min

SECONDARY OUTCOMES:
The gastric content emptying time constant [min] | up to 210 min
Area over baseline (AOB), maximum amplitude, time to maximum plasma concentration of CCK [pmol/L]. | up to 300 min
  cholecystokinin (CCK) [pmol/L].
Half emptying time from 13CO2 breath test (BT_t50) [min] | up to 300 min
Half emptying time of MRI fat volume (MRI_t50) [min] | up to 210 min
Concordance correlation of MRI fat volume MRI_t50 and breath test BT_t50 [:] | up to 300 min
Total calorie load from food consumed at the ad libitum food buffet [kcal] | up to 330 min
Amount of calories consumed from healthy foods versus unhealthy food consumed from the ad libitum food buffet [%kcal] | up to 330 min
Fatty acid concentration in gastric aspirates in percentage [%] | up to 300 min
Area over baseline (AOB), maximum amplitude, time to maximum plasma concentration of PYY [pg/mL] | up to 300 min
  peptide YY (PYY) [pg/mL]
Area over baseline (AOB), maximum amplitude, time to maximum plasma concentration of (GLP-1) [pg/mL] | up to 300 min
  glucagon-like peptide-1 (GLP-1) [pg/mL]
Area over baseline (AOB), maximum amplitude, time to maximum plasma concentration of BHB [µmol/L ] | up to 300 min
  ketone bodies β-hydroxybutyrate (BHB) [µmol/L ]
Area over baseline (AOB), maximum amplitude, time to maximum plasma concentration of triglycerides [mmol/L ] | up to 300 min
  tryglycerides [mmol/L ]

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Steingötter, PhD, Principal Investigator — University of Zurich
Locations (1):
- Division of Gastroenterology and Hepatology, University Hopsital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No